CLINICAL TRIAL: NCT04227600
Title: Phase I/II Study of JR-171 ㏌ Patients With Mucopolysaccharidosis Type I
Brief Title: A Study of JR-171 in Patients With Mucopolysaccharidosis I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JR-171-101
Record Dates: First submitted 2019-12-27; First posted 2020-01-13 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Mucopolysaccharidosis I
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part1 JR-171 (Experimental): Drug: JR-171 IV infusion, dose escalation
  Interventions: Drug: JR-171 (lepunafusp alfa)
- Part2 JR-171 (Experimental): Drug: JR-171 IV infusion, dose escalation, low dose, high dose
  Interventions: Drug: JR-171 (lepunafusp alfa)

INTERVENTIONS:
Drug: JR-171 (lepunafusp alfa) — IV infusion

SUMMARY:
Phase I/II, open-label, multicenter, multinational (Japan, Brazil and US),designed to evaluate the safety, pharmacokinetics and explore the efficacy for the treatment of mucopolysaccharidosis type I (MPS I).

DETAILED DESCRIPTION:
In the JR-171-102 study, subjects will receive either 2.0 or 4.0 mg/kg/week of JR-171 intravenously at the same dosages received at Week 12 of the JR-171-101 study.

ELIGIBILITY:
Inclusion Criteria:

* A patient aged 18 years or older in Part 1 or any age in Part 2, at the time of informed consent
* A patient from whom written informed consent can be obtained. If the patient is aged under 18 years (20 years in case of Japan) at the time of assent or willingness to participate in the study cannot be confirmed due to MPS I-related intellectual disability, informed permission from the patient's legally acceptable representative (e.g. his/her parents or guardians) need to be obtained instead of his/her consent. Even in this case, written informed consent or assent should be obtained from the patient, wherever possible
* A patient diagnosed with MPS I based on any one of the following criteria:
* Activity of IDUA enzyme below 10% of lower reference level in leucocytes or cultured skin fibroblasts, AND increased age-related urinary levels of GAGs (before enzyme replacement therapy)
* Activity of IDUA enzyme below 10% of lower reference level in leucocytes or cultured skin fibroblasts, AND presence of one pathogenic mutation in each of the alleles of the IDUA gene
* Increased age-related urinary levels of GAGs (before enzyme replacement therapy), AND presence of one pathogenic mutation in each of the alleles of the IDUA gene
* A patient diagnosed as having no or mild MPS I-related intellectual disability (able to report their own subjective symptoms) by the principal investigator or subinvestigator (Part 1 only)
* A patient who has received laronidase continuously for at least 12 weeks and has received laronidase on a stable dosage for 2 weeks immediately before the initial administration of JR-171, except for a laronidase naïve patient or a patient who has previously been treated by HSCT)
* Female patient or male patient whose co-partner is of child-bearing potential agrees to use a medically accepted, highly effective method of contraception, such as spermatocidal gel plus condom, an intrauterine device or oral contraceptives until one month after the final administration

Exclusion Criteria:

* A patient who received gene therapy treatment
* A patient who, in the opinion of the principal investigator or subinvestigator, cannot undergo lumbar puncture, including those who have a difficulty in taking a position for lumbar puncture due to joint contracture and those who are likely to develop dyspnea during lumbar puncture
* A patient who is pregnant or lactating
* A patient who has developed serious drug allergy or hypersensitivity to any drugs, in the opinion of the principal investigator or subinvestigator, is inappropriate for participation in the study
* A patient who has received another investigational product within 12 months before enrollment in the study
* A patient who, in the opinion of the principal investigator or subinvestigator, is ineligible to participate in the study out of consideration for the participant safety.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Genética e Erros Inatos do Metabolismo - IGEIM, São Paulo
- Japan (3):
  - Fukuoka Children's Hospital, Fukuoka
  - Kochi Medical School Hospital, Nankoku
  - Osaka Metropolitan University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part1, Dose-escalation: JR-171, Dose-escalation:
  * Initial dose, 0.1 mg/kg/week
  * Second dose, 1.0 mg/kg/week
  * Third dose, 2.0 mg/kg/week
  * Fourth dose, 4.0 mg/kg/week
- Part 2, Dose-escalation: JR-171, Dose-escalation:
  * Initial dose, 1.0 mg/kg/week
  * Second dose, 2.0 mg/kg/week
  * Third dose, 4.0 mg/kg/week
  * Subsequent doses, 4.0 mg/kg/week
  Participants are included as 4.0 mg/kg/week group.
- Part2, 2.0 mg: JR-171, 2.0 mg/kg/week group
- Part 2, 4.0 mg: JR-171, 4.0 mg/kg/week group
Period: Overall Study
Arm/Group | Part1, Dose-escalation | Part 2, Dose-escalation | Part2, 2.0 mg | Part 2, 4.0 mg
Started | 4 | 2 | 6 | 6
Completed | 4 | 2 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part1, Dose-escalation | Part 2, Dose-escalation | Part2, 2.0 mg | Part 2, 4.0 mg | Total
Number analyzed (Participants) | 4 | 2 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.6) | NA (NA) — Min-Max: 4-14 (since there's only two participants, only min-max data are available) Full Range data reported for the "Part 2, Dose-escalation" arm are also included in the "Total" arm. "Total" arm reflects data for all participants across all arms. | 11.0 (6.0) | 12.3 (11.4) | 19.2 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 1 | 9
  Male | 0 | 1 | 3 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 2 | 2 | 0 | 0 | 4
  Asian (Except for Japanese) | 0 | 0 | 0 | 0 | 0
  Asian (Total) | 2 | 2 | 0 | 0 | 4
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 2 | 0 | 6 | 3 | 11
  Other | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 1 | 1 | 2
  Japan | 2 | 2 | 0 | 0 | 4
  Brazil | 2 | 0 | 5 | 5 | 12
Phenotype [Count of Participants; unit: Participants]
  Hurler | 0 | 0 | 5 | 2 | 7
  Hurler-Scheie | 0 | 2 | 0 | 3 | 5
  Scheie | 4 | 0 | 1 | 1 | 6
Prior use of laronidase [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 6 | 5 | 17
  No | 0 | 0 | 0 | 1 | 1
HSCT treatment [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 1 | 0 | 1
  No | 4 | 2 | 5 | 6 | 17
Intellectual disabilities [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 5 | 4 | 10
  No | 4 | 1 | 1 | 2 | 8
Prior laronidase-related IAR [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1 | 1 | 3
  No | 3 | 2 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: Time of the first dose of JR-171 until the last visit (Week 5 for Part 1/ Week 13 for Part 2).
Population: Since participants with dose-escalation treatment continued treatment with 4.0 mg/kg/week after the first three weeks, they were analyzed as 4.0 mg/kg/week group participants
Measure: Number; unit: participants
Groups:
- Part 2, 4.0 mg: JR-171, 4.0 mg/kg/week group 4.0 mg/kg/week group includes two participants with dose-escalation treatment for the first three weeks:
  * Initial dose, 1.0 mg/kg/week
  * Second dose, 2.0 mg/kg/week
  * Third dose, 4.0 mg/kg/week
  * Subsequent doses, 4.0 mg/kg/week
Arm/Group | Part1, Dose-escalation | Part2, 2.0 mg | Part 2, 4.0 mg
Number analyzed (Participants) | 4 | 6 | 8
participants
  Adverse events | 3 | 6 | 7
  Serious adverse events | 0 | 1 | 1
  Adverse events of special interests | 1 | 3 | 3
  Adverse events leading to death | 0 | 1 | 0
  IARs (Adverse events) | 1 | 1 | 3
  Adverse drug reactions | 1 | 1 | 3
  Serious adverse drug reactions | 0 | 0 | 0
  Adverse drug reactions of special interests | 1 | 1 | 3
  Adverse drug reactions leading to death | 0 | 0 | 0
  IARs (Adverse drug reactions) | 1 | 1 | 3

2. Secondary Outcome: Pharmacokinetics of Each Dose in Part 1 (AUC0-t)
Time Frame: Week 1 to Week 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Part 1, Dose-escalation: JR-171, Dose-escalation:
  * Initial dose, 0.1 mg/kg/week
  * Second dose, 1.0 mg/kg/week
  * Third dose, 2.0 mg/kg/week
  * Fourth dose, 4.0 mg/kg/week
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
h*ng/mL
  0.1 mg/kg | 475.141 (494.371)
  1.0 mg/kg | 10293.474 (8199.941)
  2.0 mg/kg | 30776.649 (28504.162)
  4.0 mg/kg | 107077.423 (89015.623)

3. Secondary Outcome: Pharmacokinetics of Each Dose in Part 1 (Cmax)
Time Frame: Week 1 to Week 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
ng/mL
  0.1 mg/kg | 94.875 (93.331)
  1.0 mg/kg | 2825.750 (2132.838)
  2.0 mg/kg | 6889.000 (5195.335)
  4.0 mg/kg | 19040.000 (13064.037)

4. Secondary Outcome: Pharmacokinetics of Each Dose in Part 2 (AUC0-t)
Time Frame: Week 1 to Week 12
Population: There is no data for participants in dose-escalation group for plasma drug concentration after administration of JR-171.
  Though number of participants for PK set is 6 for each group, two participants from the 2.0 mg group and three participants from the 4.0 mg group was excluded from the data set since PK sample was collected by the same route as JR-171 administration and potential contamination could not be ruled out.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part2, 2.0 mg | Part 2, 4.0 mg
Number analyzed (Participants) | 4 | 3
h*ng/mL
  Week 1 | 18232.756 (9950.396) | 53691.447 (25202.412)
  Week 4 | 19466.227 (7542.104) | 33209.686 (18465.369)
  Week 12 | 22203.369 (7851.121) | 35128.134 (8312.799)

5. Secondary Outcome: Pharmacokinetics of Each Dose in Part 2 (Cmax)
Time Frame: Week 1 to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part2, 2.0 mg | Part 2, 4.0 mg
Number analyzed (Participants) | 4 | 3
ng/mL
  Week 1 | 5032.500 (2755.085) | 11526.667 (3082.229)
  Week 4 | 5421.200 (2094.819) | 8116.667 (3459.947)
  Week 12 | 6059.747 (1889.616) | 8983.333 (938.740)

6. Secondary Outcome: Heparan Sulfate Concentrations in Cerebrospinal Fluid in Part 1
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
ng/mL
  Baseline | 1131.8 (532.9)
  Week 4 | 467.0 (500.7)

7. Secondary Outcome: Dermatan Sulfate Concentrations in Cerebrospinal Fluid in Part 1
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
ng/mL
  Baseline | 264.0 (72.6)
  Week 4 | 213.0 (135.4)

8. Secondary Outcome: Heparan Sulfate Concentrations in Cerebrospinal Fluid in Part 2
Time Frame: Baseline to Week 12
Population: Since participants with dose-escalation treatment continued treatment with 4.0mg/kg/week after the first three weeks, they were analyzed as 4.0 mg/kg/group participants.
  Protocol visit was not performed at Week 12 by one participant in 4.0 mg group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part2, 2.0 mg | Part 2, 4.0 mg
Number analyzed (Participants) | 6 | 8
ng/mL
  Baseline | 3239.8 (2726.1) | 2054.0 (1542.7)
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12 | 917.5 (1216.2) | 407.6 (372.1)

9. Secondary Outcome: Dermatan Sulfate Concentrations in Cerebrospinal Fluid in Part 2
Time Frame: Baseline to Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part2, 2.0 mg | Part 2, 4.0 mg
Number analyzed (Participants) | 6 | 8
ng/mL
  Baseline | 2241.17 (2994.88) | 679.38 (451.16)
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12 | 896.80 (814.82) | 320.31 (228.30)

10. Secondary Outcome: Heparan Sulfate Concentrations in Serum in Part 1
Time Frame: Baseline to Week 5
Population: Contamination happened with Heparin or Heparin-like compounds in one participant at Week 5.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
ng/mL
  Baseline | 358.5 (52.7)
  Week 2 | 385.8 (62.5)
  Week 3 | 339.8 (59.7)
  Week 4 | 311.3 (86.3)
  Week 5: number analyzed (Participants) | 3
  Week 5 | 255.7 (67.3)

11. Secondary Outcome: Dermatan Sulfate Concentrations in Serum in Part 1
Time Frame: Baseline to Week 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
ng/mL
  Baseline | 965.0 (224.4)
  Week 2 | 929.8 (204.4)
  Week 3 | 1000.5 (200.1)
  Week 4 | 958.0 (207.1)
  Week 5 | 867.3 (241.3)

12. Secondary Outcome: Heparan Sulfate Concentrations in Serum in Part 2
Time Frame: Baseline to Week 13
Population: Participants are separated to S/H and Naive since these two will show a different trend of changes.
  Contamination happened with Heparin or Heparin-like compounds in 1 participant in 2.0 mg S/H group at W8 HS data were NA for 1 participant at W6(Not assessed), and another participant at W8, 10, 12, and 13(due to hospitalization) in 4.0 mg S/H group. Contamination happened in participant in 4.0 mg Naïve group at BL and W8, and HS data were not available at W4(due to difficult venous access).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part2, 2.0 mg Switched/HSCT: JR-171, 2.0 mg/kg/week group Participants switched treatment from laronidase or treated with allogenic HSCT before enrollment.
- Part 2, 4.0 mg Switched/HSCT: JR-171, 4.0 mg/kg/week group Participants switched treatment from laronidase or treated with allogenic HSCT before enrollment.
  4.0 mg/kg/week group includes two participants with dose-escalation treatment for the first three weeks:
  * Initial dose, 1.0 mg/kg/week
  * Second dose, 2.0 mg/kg/week
  * Third dose, 4.0 mg/kg/week
  * Subsequent doses, 4.0 mg/kg/week
- Part 2, 4.0 mg Naive: JR-171, 4.0 mg/kg/week group Participants with no treatment with laronidase or allogenic HSCT before enrollment.
Arm/Group | Part2, 2.0 mg Switched/HSCT | Part 2, 4.0 mg Switched/HSCT | Part 2, 4.0 mg Naive
Number analyzed (Participants) | 6 | 7 | 1
ng/mL
  Baseline: number analyzed (Participants) | 6 | 7 | 0
  Baseline | 668.5 (341.9) | 465.0 (314.2) |
  Week 2 | 613.3 (353.9) | 417.9 (201.0) | 1410 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 4: number analyzed (Participants) | 6 | 7 | 0
  Week 4 | 549.8 (315.9) | 368.9 (184.8) |
  Week 6: number analyzed (Participants) | 6 | 6 | 1
  Week 6 | 509.7 (331.2) | 268.3 (135.4) | 549 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 8: number analyzed (Participants) | 5 | 6 | 0
  Week 8 | 545.2 (368.2) | 265.5 (109.6) |
  Week 10: number analyzed (Participants) | 6 | 6 | 1
  Week 10 | 538.5 (357.7) | 281.3 (131.6) | 522 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 12: number analyzed (Participants) | 6 | 6 | 1
  Week 12 | 454.8 (341.2) | 274.0 (100.3) | 594 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 13: number analyzed (Participants) | 6 | 6 | 1
  Week 13 | 487.5 (306.7) | 312.8 (202.6) | 491 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.

13. Secondary Outcome: Dermatan Sulfate Concentrations in Serum in Part 2
Time Frame: Baseline to Week 13
Population: Participants are separate to S/H and Naive in this table, since these two will show a different trend of changes.
  DS data were NA for one participant at W6 (Not assessed), and for another participant at Week 8, 10, 12, and 13 (due to hospitalization) in 4.0 mg Switched/HSCT group. DS data were NA at Week 4 due to difficult venous access in participant in 4.0 mg Naïve group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part2, 2.0 mg Switched/HSCT | Part 2, 4.0 mg Switched/HSCT | Part 2, 4.0 mg Naive
Number analyzed (Participants) | 6 | 7 | 1
ng/mL
  Baseline | 1664.5 (670.8) | 1442.4 (756.6) | 4110 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 2 | 1847.5 (991.8) | 1571.6 (916.6) | 1740 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 4: number analyzed (Participants) | 6 | 7 | 0
  Week 4 | 1639.3 (792.1) | 1321.6 (687.2) |
  Week 6: number analyzed (Participants) | 6 | 6 | 1
  Week 6 | 1585.5 (686.8) | 1234.0 (807.1) | 788 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 8: number analyzed (Participants) | 6 | 6 | 1
  Week 8 | 1553.7 (811.9) | 1191.5 (681.7) | 679 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 10: number analyzed (Participants) | 6 | 6 | 1
  Week 10 | 1510.2 (704.1) | 1206.7 (719.3) | 702 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 12: number analyzed (Participants) | 6 | 6 | 1
  Week 12 | 1362.2 (642.8) | 1208.8 (763.4) | 899 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 13: number analyzed (Participants) | 6 | 6 | 1
  Week 13 | 1510.8 (699.1) | 1197.2 (811.1) | 762 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.

14. Secondary Outcome: Heparan Sulfate Concentrations in Urine in Part 1
Time Frame: Baseline to Week 5
Population: Contamination happened with Heparin or Heparin-like compounds in one participant at Week 5.
Measure: Mean (Standard Deviation); unit: µg/mgCr
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
µg/mgCr
  Baseline | 31.050 (14.339)
  Week 2 | 34.835 (11.885)
  Week 3 | 27.314 (20.634)
  Week 4 | 21.773 (19.901)
  Week 5: number analyzed (Participants) | 3
  Week 5 | 20.321 (20.612)

15. Secondary Outcome: Dermatan Sulfate Concentrations in Urine in Part 1
Time Frame: Baseline to Week 5
Measure: Mean (Standard Deviation); unit: µg/mgCr
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
µg/mgCr
  Baseline | 22.704 (13.815)
  Week 2 | 29.317 (8.615)
  Week 3 | 24.366 (16.614)
  Week 4 | 20.400 (16.880)
  Week 5 | 17.112 (17.026)

16. Secondary Outcome: Heparan Sulfate Concentrations in Urine in Part 2
Time Frame: Baseline to Week 13
Population: Participants are separated into S/H and Naive since it shows a different trend of changes.
  4 participants data were excluded from analysis due to incorrect procedure of assessment (2 each for 2.0 and 4.0 mg S/H) Data were NA for 3 participants (1 at W12 (2.0 mg)[missing creatinine data] and 1 at W6 [No assessment], 1 at W8, 10, 12, 13 (4.0 mg S/H) [due to hospitalization]) Contamination happened in participant in 4.0 mg Naïve group at BL, and HS data were NA at W2, 4, 6 (due to creatinine BLD)
Measure: Mean (Standard Deviation); unit: µg/mgCr
Arm/Group | Part2, 2.0 mg Switched/HSCT | Part 2, 4.0 mg Switched/HSCT | Part 2, 4.0 mg Naive
Number analyzed (Participants) | 4 | 5 | 1
µg/mgCr
  Baseline: number analyzed (Participants) | 4 | 5 | 0
  Baseline | 120.572 (152.114) | 35.387 (24.919) |
  Week 2: number analyzed (Participants) | 4 | 5 | 0
  Week 2 | 82.487 (103.439) | 17.962 (10.584) |
  Week 4: number analyzed (Participants) | 4 | 5 | 0
  Week 4 | 73.752 (99.221) | 10.927 (5.751) |
  Week 6: number analyzed (Participants) | 4 | 4 | 0
  Week 6 | 89.412 (122.895) | 11.662 (5.623) |
  Week 8: number analyzed (Participants) | 4 | 4 | 1
  Week 8 | 90.174 (137.086) | 6.963 (3.027) | 93.24 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 10: number analyzed (Participants) | 4 | 4 | 1
  Week 10 | 79.363 (112.278) | 9.211 (2.844) | 120.98 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 12: number analyzed (Participants) | 3 | 4 | 1
  Week 12 | 84.446 (128.037) | 10.412 (4.905) | 131.33 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 13: number analyzed (Participants) | 4 | 4 | 1
  Week 13 | 79.425 (110.272) | 15.642 (5.705) | 124.41 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.

17. Secondary Outcome: Dermatan Sulfate Concentrations in Urine in Part 2
Time Frame: Baseline to Week 13
Population: Participants are separated into S/H and Naive since it shows a different trend of changes.
  4 participants data were excluded from analysis due to incorrect procedure of assessment (2 each for 2.0 and 4.0 mg S/H) Data were NA for 3 participants (1 at W12 (2.0 mg)[missing creatinine data] and 1 at W6 [No assessment], 1 at W8, 10, 12, 13 (4.0 mg S/H) [due to hospitalization]). DS data were not available at W2, 4, and 6 (due to creatinine BLD)
Measure: Mean (Standard Deviation); unit: µg/mgCr
Arm/Group | Part2, 2.0 mg Switched/HSCT | Part 2, 4.0 mg Switched/HSCT | Part 2, 4.0 mg Naive
Number analyzed (Participants) | 4 | 5 | 1
µg/mgCr
  Baseline | 130.164 (131.983) | 39.750 (16.704) | 630.43 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 2: number analyzed (Participants) | 4 | 5 | 0
  Week 2 | 114.215 (128.204) | 30.817 (12.606) |
  Week 4: number analyzed (Participants) | 4 | 5 | 0
  Week 4 | 103.212 (117.351) | 20.873 (9.749) |
  Week 6: number analyzed (Participants) | 4 | 4 | 0
  Week 6 | 117.873 (145.111) | 20.127 (10.079) |
  Week 8: number analyzed (Participants) | 4 | 4 | 1
  Week 8 | 117.417 (158.567) | 13.330 (7.224) | 60.61 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 10: number analyzed (Participants) | 4 | 4 | 1
  Week 10 | 103.365 (124.166) | 13.171 (3.257) | 78.61 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 12: number analyzed (Participants) | 3 | 4 | 1
  Week 12 | 95.576 (131.815) | 15.406 (3.826) | 80.21 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 13: number analyzed (Participants) | 4 | 4 | 1
  Week 13 | 97.508 (116.753) | 18.432 (6.375) | 85.04 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.

18. Secondary Outcome: Liver Volumes (Body Weight Adjusted) in Part 1
Time Frame: Baseline to Week 5
Measure: Mean (Standard Deviation); unit: cm3/kg
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
cm3/kg
  Baseline | 21.912 (3.607)
  Week 5 | 22.332 (3.916)

19. Secondary Outcome: Spleen Volumes (Body Weight Adjusted) in Part 1
Time Frame: Baseline to Week 5
Measure: Mean (Standard Deviation); unit: cm3/kg
Arm/Group | Part 1, Dose-escalation
Number analyzed (Participants) | 4
cm3/kg
  Baseline | 4.342 (2.978)
  Week 5 | 4.914 (4.011)

20. Secondary Outcome: Liver Volumes (Body Weight Adjusted) in Part 2
Time Frame: Baseline to Week 13
Population: Participants are separated to Switched/HSCT and Naive in this table, since these two will show a different trend of changes.
  Liver volume data were not available for one participant each in 2.0 mg and 4.0 mg Switched/HSCT group (One couldn't arrive at the site because of the weather and another was hospitalized).
  Another participant data in 4.0 mg Switched/HSCT group was excluded from analysis since assessment was performed out of the acceptable time frame.
Measure: Mean (Standard Deviation); unit: cm3/kg
Arm/Group | Part2, 2.0 mg Switched/HSCT | Part 2, 4.0 mg Switched/HSCT | Part 2, 4.0 mg Naive
Number analyzed (Participants) | 6 | 7 | 1
cm3/kg
  Baseline | 25.027 (6.129) | 25.510 (12.295) | 35.95 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 13: number analyzed (Participants) | 5 | 5 | 1
  Week 13 | 23.795 (6.602) | 20.014 (3.778) | 29.08 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.

21. Secondary Outcome: Spleen Volumes (Body Weight Adjusted) in Part 2
Time Frame: Baseline to Week 13
Population: Participants are separated to Switched/HSCT and Naive in this table, since these two will show a different trend of changes.
  Spleen volume data were not available for one participant each in 2.0 mg and 4.0 mg Switched/HSCT group (One couldn't arrive at the site because of the weather and another was hospitalized).
  Another participant data in 4.0 mg Switched/HSCT group was excluded from analysis since assessment was performed out of the acceptable time frame.
Measure: Mean (Standard Deviation); unit: cm3/kg
Arm/Group | Part2, 2.0 mg Switched/HSCT | Part 2, 4.0 mg Switched/HSCT | Part 2, 4.0 mg Naive
Number analyzed (Participants) | 6 | 7 | 1
cm3/kg
  Baseline | 3.924 (0.766) | 4.416 (2.084) | 4.30 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.
  Week 13: number analyzed (Participants) | 5 | 5 | 1
  Week 13 | 3.629 (0.492) | 4.408 (1.486) | 3.10 (NA) — Since the group has one participant, the value in Mean is not a mean value but the actual measured value for the participant.

ADVERSE EVENTS:
Time Frame: Time of the first dose of JR-171 until the last visit (Week 5 for Part 1/ Week 13 for Part 2). Events occurring within 28 days after the time of observation at Week 5 in Part 1/Week 13 in Part 2 or discontinuation that are considered related to JR-171 will also be collected.
Groups:
- Part1, Dose-escalation: JR-171, Dose-escalation:
  * Initial administration, 0.1 mg/kg/week
  * Second administration, 1.0 mg/kg/week
  * Third administration, 2.0 mg/kg/week
  * Fourth administration, 4.0 mg/kg/week
- Part 2, 4.0 mg: JR-171, 4.0 mg/kg/week group 4.0 mg/kg/week group includes two participants with dose-escalation treatment for the first three weeks:
  * Initial dose, 1.0 mg/kg/week
  * Second dose, 2.0 mg/kg/week
  * Third dose, 4.0 mg/kg/week
  * Subsequent doses, 4.0 mg/kg/week
  Since participants with dose-escalation treatment continued treatment with 4.0mg/kg/week after the first three weeks, they were analyzed as 4.0 mg/kg/group participants.
Arm/Group | Part1, Dose-escalation | Part2, 2.0 mg | Part 2, 4.0 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 1/8
Other Adverse Events (participants affected / at risk) | 3/4 | 6/6 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1, Dose-escalation (N=4) | Part2, 2.0 mg (N=6) | Part 2, 4.0 mg (N=8)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1, Dose-escalation (N=4) | Part2, 2.0 mg (N=6) | Part 2, 4.0 mg (N=8)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cutaneous larva migrans (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (4)
Blood iron decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
CSF pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte morphology abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04227600/Prot_SAP_002.pdf